CLINICAL TRIAL: NCT00768872
Title: Neuro Ambulatory Data Recorder (ADR) Spinal Cord Stimulation (SCS) Study
Brief Title: Spinal Cord Stimulation Research Study
Acronym: ADR-SCS
Status: Completed | Type: Observational
Sponsor: MedtronicNeuro (Industry)
Responsible Party: Sponsor
Other Study IDs: 1644
Record Dates: First submitted 2008-10-07; First posted 2008-10-08 (Estimated); Last update posted 2016-10-14 (Estimated); Status verified 2016-10

CONDITIONS: Chronic Low Back and Leg Pain
Keywords: activity, spinal cord stimulation, pain
MeSH Terms: conditions — Motor Activity; Pain

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to characterize a patient's activity levels before and after spinal cord stimulation therapy.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Candidate for SCS device trial
* Subject is ambulatory
* Diagnosed with low back pain or low back pain plus leg pain for at least 6 months
* Undergoing treatment for low back pain or low back pain plus leg pain
* Does not have or has not had a previous SCS implant
* Willing and able to complete protocol requirements
* Willing and able to sign the study-specific Informed Consent form
* Male or non-pregnant female

Exclusion Criteria:

* Have plans to enroll in another clinical study during their participation in this study, or are currently enrolled in a clinical study that could interfere in participation in the trial or affect the scientific soundness of this study
* Cancer or any other malignant disease
* Present or past diagnosis of schizophrenia or of delusional, psychotic, or dissociative disorder
* A pain-related surgery in the previous 12 weeks of enrollment, the intent to undergo surgery during the period of the study
* Non-English speaking or an inability to complete questionnaires accurately

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Candidates for Spinal Cord Stimulation
Sampling Method: Non-Probability Sample
Enrollment: 66 (Actual)
Dates: Start 2008-10; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in Physical Activity (total centi-Gs per 5.125 seconds) | 4, 12, 24 weeks post implant
Change from Baseline in Posture Parameters (minutes per 24 hours) | 4, 12, 24 weeks post implant

CONTACTS AND LOCATIONS:
Overall Officials: David M Schultz, MD, Principal Investigator — Medical Advanced Pain Specialists (MAPS); Robert Jamison, Ph.D, Principal Investigator — Brigham and Women's Hospital; Eric Grigsby, M.D., Principal Investigator — Napa Pain Institute
Locations (3):
- United States (3):
  - Napa Pain Institute, Napa, California
  - Brigham and Women's Hospital, Chestnut Hill, Massachusetts
  - Medical Advanced Pain Specialists (MAPS), Edina, Minnesota